CLINICAL TRIAL: NCT02593110
Title: Telmisartan Plus Exercise to Improve Functioning in Peripheral Artery Disease
Acronym: TELEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Mary McDermott, Jeremiah Stamler Professor, Northwestern University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU00200954; R01HL126117 (NIH)
Record Dates: First submitted 2015-10-27; First posted 2015-10-30 (Estimated); Results first posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-12

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Telmisartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Telmisartan + Supervised Treadmill Exercise Therapy (Active Comparator): Participants in this group will receive both daily telmisartan and supervised treadmill exercise three days weekly for six months.
  Interventions: Behavioral: Supervised Treadmill Exercise Therapy; Drug: Telmisartan
- Telmisartan + "No Exercise" Control Group (Active Comparator): Participants in this group will receive daily telmisartan and attend weekly educational lectures at the medical center for six months.
  Interventions: Drug: Telmisartan; Other: "No exercise" control group
- Placebo + Supervised Treadmill Exercise Therapy (Active Comparator): Participants randomized to this group will receive daily placebo and supervised treadmill exercise three times weekly for six months.
  Interventions: Behavioral: Supervised Treadmill Exercise Therapy; Drug: Placebo
- Placebo + "No Exercise" Control Group (Placebo Comparator): Participants randomized to this group will receive daily placebo and health education lectures weekly for six months.
  Interventions: Other: "No exercise" control group; Drug: Placebo

INTERVENTIONS:
Behavioral: Supervised Treadmill Exercise Therapy — Participants randomized to the exercise intervention will receive supervised treadmill exercise three times weekly for six months.
  Other Names: Treadmill exercise
  Arms: Placebo + Supervised Treadmill Exercise Therapy; Telmisartan + Supervised Treadmill Exercise Therapy
Drug: Telmisartan — Participants randomized to the telmisartan arm of the study will take 20 mg or 40 mg of telmisartan daily based on the results of their study run-in. Participants will have their dose increased to up to 80 mg as tolerated.
  Other Names: Micardis
  Arms: Telmisartan + "No Exercise" Control Group; Telmisartan + Supervised Treadmill Exercise Therapy
Other: "No exercise" control group — Participants randomized to the attention control group will attend weekly one-hour educational sessions at Northwestern University for six months.
  Other Names: Attention control group
  Arms: Placebo + "No Exercise" Control Group; Telmisartan + "No Exercise" Control Group
Drug: Placebo
  Arms: Placebo + "No Exercise" Control Group; Placebo + Supervised Treadmill Exercise Therapy

SUMMARY:
The TELEX trial will establish whether telmisartan alone improves walking performance in people with peripheral artery disease (PAD). The TELEX trial will also determine whether telmisartan plus supervised exercise improves walking performance more than either therapy alone. TELEX is a randomized controlled clinical trial (2 x 2 factorial design) of 112 participants with PAD randomized to one of four arms: Group A: telmisartan + supervised exercise therapy; Group B: telmisartan + a "no exercise" control group; Group C: placebo + supervised exercise therapy; and Group D: placebo + a "no exercise" control group.

ELIGIBILITY:
Inclusion Criteria:

All participants will have PAD. PAD will be defined as follows. First, an ABI <= 0.90 at the baseline study visit is an inclusion criterion for PAD. Second, potential participants who have an ABI > 0.90 but ≤ 1.00 and experience a 20% or higher drop in ABI after heel-rise exercise will be eligible. Third, potential participants with an ABI > 0.90 who have vascular lab evidence of PAD or angiographic evidence of PAD will be eligible. Finally, potential participants with a history of lower extremity revascularization who do not meet the criterion above and have an ABI > 0.90 with a 20% or higher drop in ABI after heel-rise exercise will be eligible.

Exclusion Criteria:

1. Above or below knee amputation, critical limb ischemia, wheelchair confinement, inability to walk without a walker, or current foot ulcer.
2. Walking is limited by a condition other than PAD.
3. > Class II NYHA heart failure or angina, increase in angina, angina at rest, or abnormal baseline treadmill stress test. Potential participants may become eligible following an abnormal baseline treadmill stress test if they have evidence of an absence of coronary ischemia based on testing with their own physician.
4. Currently taking an angiotensin receptor blocker or an ACE inhibitor or use of these medications in the past three months.
5. Currently taking aliskiren (Tekturna).
6. Blood pressure < 100/50 at baseline or potassium > 5.0 meq/L at baseline.
7. Blood pressure < 100/50 after run-in or potassium >= 5.5 meq/L at the end of run-in.
8. Severe hepatic impairment defined by two or more liver function enzyme values greater than 2.5 the upper limit of normal.
9. Acute decline in renal function on telmisartan, defined as a 30% or greater decline in eGFR following the two-week run-in as compared to baseline. If the participant had a baseline eGFR performed by his/her physician within two months of the baseline eGFR for the TELEX trial, the participant's physician's eGFR may be considered the baseline measure, at the study principal investigator's discretion.
10. Allergy to ARBs.
11. Failure to successfully complete the 2-week study run-in, defined as failing to attend the health education and treadmill exercise run-in sessions and/or failing to take the study medication daily for 10 or more days in the two-week period (i.e. one pill per day for > 10 days out of the 14 day run-in period).
12. Surgery including lower extremity revascularization, coronary revascularization with stenting, or orthopedic surgery during the past 3 months or anticipated in the next 6 months or myocardial infarction or stroke in the past 3 months.
13. Major medical illness including renal disease requiring dialysis, lung disease requiring oxygen, Parkinson's disease, a life-threatening illness with life expectancy less than six months, or cancer requiring treatment in the previous two years. [NOTE: potential participants may still qualify if they have had treatment for an early stage cancer in the past two years and the prognosis is excellent. Participants who only use oxygen at night may still qualify.]
14. MMSE score < 23 or dementia.
15. Currently walking regularly for exercise at a level similar to the study intervention.
16. Participation in another clinical trial or cardiac rehabilitation or completion of a clinical trial or cardiac rehabilitation in the previous three months. [NOTE: after completing a stem cell or gene therapy intervention, participants will become eligible after the final study follow-up visit of the stem cell or gene therapy study so long as at least six months have passed since the final intervention administration. After completing an exercise intervention or a supplement or drug therapy (other than stem cell or gene therapy), participants will be eligible after the final study follow-up visit as long as at least three months have passed since the final intervention of the trial.]
17. Non-English speaking, a visual impairment that limits walking ability, or a hearing impairment that interferes with study participation.
18. Congestive heart failure with an ejection fraction <40.
19. In addition to the above criteria, investigator discretion will be used to determine if the trial is unsafe or not a good fit for the potential participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2016-01-04 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary McDermott, MD, Principal Investigator — Northwestern University
Locations (3):
- United States (3):
  - Northwestern University, Chicago, Illinois
  - Tulane University, New Orleans, Louisiana
  - Ochsner Medical Center, New Orleans, Louisiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McDermott MM, Bazzano L, Peterson CA, Sufit R, Ferrucci L, Domanchuk K, Zhao L, Polonsky TS, Zhang D, Lloyd-Jones D, Leeuwenburgh C, Guralnik JM, Kibbe MR, Kosmac K, Criqui MH, Tian L. Effect of Telmisartan on Walking Performance in Patients With Lower Extremity Peripheral Artery Disease: The TELEX Randomized Clinical Trial. JAMA. 2022 Oct 4;328(13):1315-1325. doi: 10.1001/jama.2022.16797. PMID 36194220

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo + Supervised Treadmill Exercise Therapy: Participants randomized to this group will receive daily placebo and supervised treadmill exercise three times weekly for six months.
  Supervised Treadmill Exercise Therapy: Participants randomized to the exercise intervention will receive supervised treadmill exercise three times weekly for six months.
  Placebo
- Placebo + "No Exercise" Control Group: Participants randomized to this group will receive daily placebo and health education lectures weekly for six months.
  "No exercise" control group: Participants randomized to the attention control group will attend weekly one-hour educational sessions at Northwestern University for six months.
  Placebo
Period: Overall Study
Arm/Group | Telmisartan + Supervised Treadmill Exercise Therapy | Telmisartan + "No Exercise" Control Group | Placebo + Supervised Treadmill Exercise Therapy | Placebo + "No Exercise" Control Group
Started | 30 | 29 | 28 | 27
Completed | 30 | 26 | 24 | 25
Not Completed | 0 | 3 | 4 | 2
Not completed — Withdrawal by Subject | 0 | 3 | 3 | 2
Not completed — Death | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telmisartan + Supervised Treadmill Exercise Therapy | Telmisartan + "No Exercise" Control Group | Placebo + Supervised Treadmill Exercise Therapy | Placebo + "No Exercise" Control Group | Total
Number analyzed (Participants) | 30 | 29 | 28 | 27 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.5 (8.9) | 66.9 (10.0) | 65.8 (9.4) | 67.9 (11.5) | 67.3 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 15 | 9 | 46
  Male | 18 | 19 | 13 | 18 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 2 | 1 | 7
  Not Hispanic or Latino | 27 | 23 | 26 | 26 | 102
  Unknown or Not Reported | 2 | 3 | 0 | 0 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 22 | 21 | 18 | 20 | 81
  White | 6 | 5 | 9 | 6 | 26
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 1 | 1 | 5
Ankle-brachial index [Mean (Standard Deviation); unit: ratio] — ABI is a ratio of Doppler recorded arm and ankle pressures and that a value < 0.90 indicates PAD
  ratio | 0.67 (0.23) | 0.77 (0.30) | 0.78 (0.23) | 0.69 (0.17) | 0.73 (0.24)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 30.45 (7.49) | 27.61 (6.23) | 28.73 (6.40) | 28.20 (5.75) | 28.77 (6.53)
Six-min walk distance [Mean (Standard Deviation); unit: meters] | 327.30 (96.58) | 359.62 (84.41) | 317.42 (123.31) | 374.55 (122.40) | 344.29 (108.51)

OUTCOME MEASURES:

1. Primary Outcome: Six-minute Walk Performance
Description: We will determine whether telmisartan therapy with or without exercise improves six-minute walk distance at 6-month follow-up, compared to placebo with or without exercise (i.e. two group comparisons of all participants randomized to telmisartan vs. all participants randomized to placebo).
Time Frame: Change from baseline to six-month follow-up
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Telmisartan + Supervised Treadmill Exercise Therapy | Telmisartan + "No Exercise" Control Group | Placebo + Supervised Treadmill Exercise Therapy | Placebo + "No Exercise" Control Group
Number analyzed (Participants) | 30 | 25 | 23 | 24
meters | 5.86 (67.21) | -3.92 (47.33) | 30.27 (29.44) | -4.62 (42.54)
Statistical Analysis 1: Comparison: Telmisartan + Supervised Treadmill Exercise Therapy vs Placebo + Supervised Treadmill Exercise Therapy; Test type: Superiority; p = 0.1107, ANCOVA; Mean Difference (Final Values) = -24.41, 95% CI 2-sided [-54.59 to 5.78]
Statistical Analysis 2: Comparison: Telmisartan + Supervised Treadmill Exercise Therapy vs Telmisartan + "No Exercise" Control Group; Test type: Superiority; p = 0.5378, ANCOVA; Mean Difference (Final Values) = 9.78, 95% CI 2-sided [-21.84 to 41.39]
Statistical Analysis 3: Comparison: Telmisartan + "No Exercise" Control Group vs Placebo + "No Exercise" Control Group; Test type: Superiority; p = 0.9560, ANCOVA; Mean Difference (Final Values) = 0.71, 95% CI 2-sided [-24.96 to 26.38]

2. Secondary Outcome: Maximal Treadmill Walking Distance
Description: In the treadmill walking test, participants walk on either a gardner or modified gardner protocol until they stop the test. Distance walked is recorded.
Time Frame: Change from baseline to six-month follow-up
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Telmisartan + Supervised Treadmill Exercise Therapy | Telmisartan + "No Exercise" Control Group | Placebo + Supervised Treadmill Exercise Therapy | Placebo + "No Exercise" Control Group
Number analyzed (Participants) | 26 | 24 | 19 | 20
meters | 207.99 (150.44) | 66.21 (226.81) | 176.64 (259.51) | 80.96 (178.73)
Statistical Analysis 1: Comparison: Telmisartan + Supervised Treadmill Exercise Therapy vs Placebo + Supervised Treadmill Exercise Therapy; Test type: Superiority; p = 0.6121, ANCOVA; Mean Difference (Final Values) = 31.35, 95% CI 2-sided [-92.42 to 155.12]
Statistical Analysis 2: Comparison: Telmisartan + Supervised Treadmill Exercise Therapy vs Telmisartan + "No Exercise" Control Group; Test type: Superiority; p = 0.0116, ANCOVA; Mean Difference (Final Values) = 141.78, 95% CI 2-sided [33.14 to 250.42]
Statistical Analysis 3: Comparison: Telmisartan + "No Exercise" Control Group vs Placebo + "No Exercise" Control Group; Test type: Superiority; p = 0.8146, ANCOVA; Mean Difference (Final Values) = -14.75, 95% CI 2-sided [-140.89 to 111.39]

3. Secondary Outcome: Walking Impairment Questionnaire (WIQ) Distance Score
Description: The WIQ is a well validated questionnaire that measures patient-reported walking limitations in distance and speed and stair-climbing. They are scored on a 0-100 scale and that 100 indicates the best possible score.
Time Frame: Change from baseline to six-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telmisartan + Supervised Treadmill Exercise Therapy | Telmisartan + "No Exercise" Control Group | Placebo + Supervised Treadmill Exercise Therapy | Placebo + "No Exercise" Control Group
Number analyzed (Participants) | 29 | 26 | 24 | 24
score on a scale | 8.77 (26.35) | 6.33 (33.69) | 7.85 (12.42) | -0.55 (17.91)
Statistical Analysis 1: Comparison: Telmisartan + Supervised Treadmill Exercise Therapy vs Placebo + Supervised Treadmill Exercise Therapy; Test type: Superiority; p = 0.8755, ANCOVA; Mean Difference (Final Values) = 0.92, 95% CI 2-sided [-10.84 to 12.68]
Statistical Analysis 2: Comparison: Telmisartan + Supervised Treadmill Exercise Therapy vs Telmisartan + "No Exercise" Control Group; Test type: Superiority; p = 0.7651, ANCOVA; Mean Difference (Final Values) = 2.44, 95% CI 2-sided [-13.83 to 18.70]
Statistical Analysis 3: Comparison: Telmisartan + "No Exercise" Control Group vs Placebo + "No Exercise" Control Group; Test type: Superiority; p = 0.3776, ANCOVA; Mean Difference (Final Values) = 6.88, 95% CI 2-sided [-8.65 to 22.41]

4. Secondary Outcome: SF-36 Physical Functioning Score
Description: The SF-36 physical functioning score will be used to measure quality of life. They are scored on a 0-100 scale and that 100 indicates the best possible score.
Time Frame: Change from baseline to six-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telmisartan + Supervised Treadmill Exercise Therapy | Telmisartan + "No Exercise" Control Group | Placebo + Supervised Treadmill Exercise Therapy | Placebo + "No Exercise" Control Group
Number analyzed (Participants) | 29 | 26 | 24 | 24
score on a scale | 0.69 (21.16) | 5.96 (20.69) | 8.75 (21.68) | 0.21 (20.56)
Statistical Analysis 1: Comparison: Telmisartan + Supervised Treadmill Exercise Therapy vs Placebo + Supervised Treadmill Exercise Therapy; Test type: Superiority; p = 0.1782, ANCOVA; Mean Difference (Final Values) = -8.06, 95% CI 2-sided [-19.91 to 3.79]
Statistical Analysis 2: Comparison: Telmisartan + Supervised Treadmill Exercise Therapy vs Telmisartan + "No Exercise" Control Group; Test type: Superiority; p = 0.3555, ANCOVA; Mean Difference (Final Values) = -5.27, 95% CI 2-sided [-16.61 to 6.07]
Statistical Analysis 3: Comparison: Telmisartan + "No Exercise" Control Group vs Placebo + "No Exercise" Control Group; Test type: Superiority; p = 0.3294, ANCOVA; Mean Difference (Final Values) = 5.75, 95% CI 2-sided [-5.99 to 17.49]

5. Secondary Outcome: Walking Impairment Questionnaire (WIQ) Speed Score
Description: as for outcome 3
Time Frame: Change from baseline to six-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telmisartan + Supervised Treadmill Exercise Therapy | Telmisartan + "No Exercise" Control Group | Placebo + Supervised Treadmill Exercise Therapy | Placebo + "No Exercise" Control Group
Number analyzed (Participants) | 29 | 26 | 24 | 24
score on a scale | 2.74 (25.64) | 4.81 (26.41) | 11.46 (16.52) | 1.72 (17.36)
Statistical Analysis 1: Comparison: Telmisartan + Supervised Treadmill Exercise Therapy vs Placebo + Supervised Treadmill Exercise Therapy; Test type: Superiority; p = 0.1569, ANCOVA; Mean Difference (Final Values) = -8.72, 95% CI 2-sided [-20.91 to 3.47]
Statistical Analysis 2: Comparison: Telmisartan + Supervised Treadmill Exercise Therapy vs Telmisartan + "No Exercise" Control Group; Test type: Superiority; p = 0.7692, ANCOVA; Mean Difference (Final Values) = -2.07, 95% CI 2-sided [-16.16 to 12.02]
Statistical Analysis 3: Comparison: Telmisartan + "No Exercise" Control Group vs Placebo + "No Exercise" Control Group; Test type: Superiority; p = 0.6306, ANCOVA; Mean Difference (Final Values) = 3.09, 95% CI 2-sided [-9.74 to 15.91]

6. Secondary Outcome: Walking Impairment Questionnaire (WIQ) Stair-climbing Score
Description: as for outcome 3
Time Frame: Change from baseline to six-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telmisartan + Supervised Treadmill Exercise Therapy | Telmisartan + "No Exercise" Control Group | Placebo + Supervised Treadmill Exercise Therapy | Placebo + "No Exercise" Control Group
Number analyzed (Participants) | 29 | 26 | 24 | 24
score on a scale | 2.73 (34.81) | 3.37 (28.58) | 10.59 (24.14) | -2.08 (21.21)
Statistical Analysis 1: Comparison: Telmisartan + Supervised Treadmill Exercise Therapy vs Placebo + Supervised Treadmill Exercise Therapy; Test type: Superiority; p = 0.3542, ANCOVA; Mean Difference (Final Values) = -7.86, 95% CI 2-sided [-24.74 to 9.02]
Statistical Analysis 2: Comparison: Telmisartan + Supervised Treadmill Exercise Therapy vs Telmisartan + "No Exercise" Control Group; Test type: Superiority; p = 0.9417, ANCOVA; Mean Difference (Final Values) = -0.64, 95% CI 2-sided [-17.98 to 16.71]
Statistical Analysis 3: Comparison: Telmisartan + "No Exercise" Control Group vs Placebo + "No Exercise" Control Group; Test type: Superiority; p = 0.4508, ANCOVA; Mean Difference (Final Values) = 5.45, 95% CI 2-sided [-8.96 to 19.86]

ADVERSE EVENTS:
Time Frame: Adverse events data were collected during the 6-month intervention period.
Arm/Group | Telmisartan + Supervised Treadmill Exercise Therapy | Telmisartan + "No Exercise" Control Group | Placebo + Supervised Treadmill Exercise Therapy | Placebo + "No Exercise" Control Group
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/29 | 1/28 | 0/27
Serious Adverse Events (participants affected / at risk) | 4/30 | 5/29 | 6/28 | 7/27
Other Adverse Events (participants affected / at risk) | 20/30 | 15/29 | 23/28 | 18/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telmisartan + Supervised Treadmill Exercise Therapy (N=30) | Telmisartan + "No Exercise" Control Group (N=29) | Placebo + Supervised Treadmill Exercise Therapy (N=28) | Placebo + "No Exercise" Control Group (N=27)
Depression (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Coronary revascularization (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lower extremity revascularization (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Stroke (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Toe gangrene/infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anemia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic aneurysm (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carotid artery revascularization (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain- non-cardiac (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Elective orthopedic surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Elective pacemaker placement (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hematoma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertensive urgency (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower extremity revascularization/Amputation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Opioid addiction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Panic attack (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toe infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telmisartan + Supervised Treadmill Exercise Therapy (N=30) | Telmisartan + "No Exercise" Control Group (N=29) | Placebo + Supervised Treadmill Exercise Therapy (N=28) | Placebo + "No Exercise" Control Group (N=27)
Increase in shortness of breath (General disorders) | 7 (11) | 9 (16) | 7 (13) | 10 (14)
New chest pain during exertion (General disorders) | 2 (5) | 4 (4) | 3 (3) | 2 (2)
Sinus discomfort or congestion (General disorders) | 20 (54) | 14 (46) | 16 (50) | 18 (60)
Back pain (General disorders) | 18 (74) | 15 (54) | 23 (85) | 15 (60)
Diarrhea (General disorders) | 17 (37) | 14 (38) | 17 (61) | 11 (33)
Dizziness or lightheadedness (General disorders) | 9 (14) | 9 (15) | 9 (12) | 8 (14)
Swelling in the face, lips or tongue (General disorders) | 5 (10) | 1 (2) | 2 (2) | 1 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-07): https://cdn.clinicaltrials.gov/large-docs/10/NCT02593110/Prot_SAP_000.pdf